CLINICAL TRIAL: NCT03422341
Title: Prospective Study for Clinical Validation of the Molecular-Based GenePOC Strep A, C/G Assay for the Detection and Identification of Group A β-hemolytic Streptococcus (Streptococcus Pyogenes) and Pyogenic Group C and G β-hemolytic Streptococcus (Streptococcus Dysgalactiae Subsp. Equisimilis) Nucleic Acids From Throat Swab Samples Obtained From Patients With Signs and Symptoms of Pharyngitis.
Brief Title: Validation of the GenePOC Strep A, C/G Assay for Detecting Group A, C and G β-hemolytic Streptococcus From Throat Swabs.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GPC03-002
Record Dates: First submitted 2018-01-23; First posted 2018-02-05 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2019-06

CONDITIONS: Pharyngitis, Infective
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- GenePOC testing (Experimental): The swab will be used for the testing on the revogene using the GenePOC Strep A, C/G assay.
  Intervention will be the Comparison between GenePOC CR and Reference Method.
  Interventions: Device: Comparison between GenePOC CR and Reference Method
- Reference Method (Active Comparator): The swab will be used to detect the presence or absence of Strep A, C/G using standard microbiology method.
  Intervention will be the Comparison between GenePOC CR and Reference Method.
  Interventions: Device: Comparison between GenePOC CR and Reference Method

INTERVENTIONS:
Device: Comparison between GenePOC CR and Reference Method — The collected swab will be tested with both the GenePOC Strep A, C/G assay and the Reference Method defined as standard microbiology culture and strain identification using a MALDI TOF.

SUMMARY:
The primary purpose of this clinical investigation is to establish the performance of the GenePOC Strep A, C/G assay on the revogene. This will be achieved by comparing the test to a conventional method for detection of Group A β-hemolytic Streptococcus (GAS) and pyogenic Group C and G β-hemolytic Streptococcus (GCS/GGS) in throat swab samples.

DETAILED DESCRIPTION:
The GenePOC Strep A, C/G assay will be performed using the revogene™ instrument. The revogene instrument, used in conjunction with appropriate reagents, is capable of automated cell lysis, dilution of nucleic acids from multiple sample types as well as automated amplification and detection of target nucleic acid sequences.

A dual swab sample is collected when ICF is signed by patient. One of the swab will be tested on the revogene™, and the second swab will be tested with standard microbiology method at a Reference Center.

ELIGIBILITY:
Inclusion Criteria:

* Samples from patients suspected of having signs and symptoms of a pharyngitis infection
* Patient that signed the approved Informed Consent Form (if applicable)
* Patient older than 2 years of age
* Only one (1) compliant sample per patient is allowed
* Use of dual swab with either liquid Stuart or liquid Amies transport Medium

Exclusion Criteria:

• Patient/sample not meeting inclusion criteria above

Min Age: 25 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 497 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

PRIMARY OUTCOMES:
Performance characteristics of the GenePOC Streap A, C/G assay | Up to 14 months
  To establish the performance characteristics of the GenePOC Strep A, C/G assay for its use in determining the presence of Strep A, C/G in throat swab samples obtained from patients with signs and symptoms of pharyngitis infection.
  * Sensitivity will be estimated as the proportion of positives that are correctly identified by the GenePOC Strep A, C/G assay when compared to the Reference Method.
  * Specificity will be established as the proportion of negatives that are correctly identified by the GenePOC Strep A, C/G assay when compared to the Reference Method.

SECONDARY OUTCOMES:
Positive and Negative Predictive Values (PPV and NPV) | Up to 14 months
  To establish the Positive and Negative Predictive Values (PPV and NPV) of the GenePOC Strep A, C/G assay.
  PPV will be calculated as the proportion of positive results with the GenePOC Strep A, C/G assay that are true positive results when compared to the Reference Method.
  NPV will be calculated as the proportion of negative results with the GenePOC Strep A, C/G assay that are true negative results when compared to the Reference Method.
Unresolved sample results | Up to 14 months
  To establish the rate of unresolved results for the GenePOC Strep A, C/G assay due to sample processing control failure (unresolved sample results).
Indeterminate sample results | Up to 14 months
  To establish the rate of indeterminate results for the GenePOC Strep A, C/G assay due to an instrument failure (indeterminate results).

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Allibert, Study Director — Meridian Bioscience, Inc.
Locations (8):
- United States (5):
  - Valley Children's Hospital, Madera, California
  - Wishard Health Services, Indianapolis, Indiana
  - Detroit Medical Center University Laboratories, Detroit, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - BC Children's and Women's Hospital, Vancouver, British Columbia
  - Mount Sinai Services, Toronto, Ontario
  - Centre de Recherche Saint-Louis, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No